CLINICAL TRIAL: NCT04801238
Title: preGallstep: One-step Laparoscopic Cholecystectomy, Common Bile Duct Exploration and Stone Extraction Versus Two-step Endoscopic Retrograde Cholangiography and Stone Extraction Plus Laparoscopic Cholecystectomy for Common Bile Duct Stones
Brief Title: preGallstep - A Clinical Pilot Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lars Tue Sorensen (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other)
Responsible Party: Sponsor-Investigator, Lars Tue Sorensen, Head of Surgical Department, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: preGallstep
Record Dates: First submitted 2021-03-08; First posted 2021-03-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Pancreatitis; Cholangitis; Cholecystitis; Gallstone; Jaundice, Obstructive
Keywords: Obstructive Jaundice; gallbladder stones; common bile duct; ERC; LCBDE; Laparoscopic; Cholecystectomy
MeSH Terms: conditions — Pancreatitis; Cholangitis; Cholecystitis; Gallstones; Jaundice, Obstructive; Cholecystolithiasis

STUDY DESIGN:
Intervention Model Description: The preGallStep is an investigator-initiated, multicentre randomised parallel group, clinical pilot trial, with blinded outcome assessment investigating one-step laparoscopic cholecystectomy with common bile duct exploration and stone extraction versus two-step endoscopic retrograde cholangiography with stone extraction plus laparoscopic cholecystectomy for patients with common bile duct stones.
Who Masked: Outcomes Assessor
Masking Description: The obvious advantages of a one-step procedure compared with a two-step procedure are the fewer surgical procedures required to clear CBDS and to remove the gallbladder. Due to the nature of the surgical interventions, blinding of patients or physicians is not possible for this trial. Most of the outcomes are dependent on the physician's clinical assessment. However, we will engage a blinded adjudication committee of 3 independent experts who will examine medical charts from randomisation to 90-day follow-up for outcome assessment. Photocopies of the medical charts will have intervention blinded. Also photocopies or print outs of medical charts will be changed so that follow up interventions will become blinded for initial intervention in both intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCBDE + LC (Active Comparator): Laparoscopic common bile duct exploration with laparoscopic cholecystectomy
  Interventions: Procedure: LCBDE + LC
- ERC + LC (Active Comparator): Endoscopic retrograde cholangiography with laparoscopic cholecystectomy
  Interventions: Procedure: ERC + LC

INTERVENTIONS:
Procedure: LCBDE + LC — Experimental group: Laparoscopic common bile duct exploration (LCBDE) + laparoscopic cholecystectomy (LC) is performed under full anaesthesia. Once the dissection has exposed the cystic a clip or ligature is placed peripherally on the cystic duct. Through an incision in the duct central to the clip or ligature a cholangiogram catheter is introduced into the cystic duct and the cholangiogram is completed.
  After identification of the bile duct stones and anatomy, a cholangioscope is introduced through the duct incision into common bile duct. The stones are identified visually and removed by Dormia basket. If the stones are very large, they may be partitioned mechanically or by electrohydraulic lithotripsy. In the presence of CBDS wedged in the papilla these stones will be removed and a secondary cholangiogram will be performed. Subsequently, the cholangioscope is taken out. Then the cystic duct is divided and the gallbladder is dissected out from the liver by hook cautery and removed.
  Arms: LCBDE + LC
Procedure: ERC + LC — Control intervention: (First step) Endoscopic retrograde cholangiography (ERC) is routinely performed in sedation but or in full anaesthesia. ERC is performed with the patient in the supine position. The endoscope is passed down to the second part of the duodenum where the papilla is identified. Cannulation of the papilla and the common bile duct is performed with a papillotome and a guidewire. A cholangiography will confirm the presence, location and size of the CBDS and aims in further choice of extraction method. Stones can be extracted by papillotomy and by either balloon or by a basket. Additional balloon dilation of the papilla, or lithotripsy may be required. If stone extraction is incomplete or if the conditions are unclear a temporary common bile duct stent is placed which has to be removed with additional ERC after 1-2 months (Second step) laparoscopic cholecystectomy is performed after 2-14 days
  Arms: ERC + LC

SUMMARY:
In Denmark, more than 7500 cholecystectomies are performed every year. Common bile duct gallstones (CBDS) are found in 3.4% to 18% of patients undergoing cholecystectomy. A two-step approach including endoscopic retrograde cholangiography (ERC) with stone extraction and papillotomy with subsequent laparoscopic cholecystectomy has become gold standard for treatment of CBDS in Denmark. However, ERC is associated with a high risk of complications and more than 50% of patients require multiple ERCs. Recent meta analyses find that a one-step approach might be superior in terms of safety, CBDS clearance rate, hospital stay, operative time, hospital cost and stone recurrence, but much more data is needed.

The preGallstep trial is an investigator-initiated multicentre randomised clinical pilot trial with blinded outcome assessment investigating a novel one-step laparoscopic cholecystectomy with common bile duct exploration and stone extraction versus conventional two-step endoscopic retrograde cholangiography with stone extraction plus a subsequent laparoscopic cholecystectomy for patients with CBDS. After enrolment, the participant will be randomised to one of the two treatment approaches. Adult patients with imaging confirmed CBDS are eligible for inclusion. Potential postoperative complications will be assessed within 90 days following the procedure.

The primary outcome is the proportion of serious adverse events (corresponding to a Clavien-Dindo score II or above) requiring re-intervention within 90 days of the initial procedure. This outcome will be used for a future sample size calculation. The sample size estimate, the inclusion rate and the estimated length of subsequent trial will be used to determine the feasibility of a large pragmatic and confirmatory trial.

We hypothesize that the one-step approach will significantly reduce the risk of complications and number of treatments needed thereby making a difference to hundreds of people in Denmark each year.

DETAILED DESCRIPTION:
Purpose The preGallstep pilot trial is a pilot randomised clinical trial investigating two different surgical methods in patients with common bile duct stones: one-step laparoscopic cholecystectomy with common bile duct exploration (experimental intervention) versus two-step endoscopic retrograde cholangiography with stone extraction plus subsequent laparoscopic cholecystectomy (control intervention) for the removal of common bile duct stones.

The investigators alternative hypothesis is that both patient safety, assessed by serious adverse events, as well as the number of procedures needed to obtain stone clearance are better in the one-step approach than in the control approach. However, based on updated systematic review of previously conducted randomised clinical trials (RCTs) the investigators are not able to say which procedure is preferable. Further analysis of these previous RTCs show they are very far from obtaining a confirmatory sample size, thus illustrating the need for larger multicenter trials.

Prior to conducting a large pragmatic and confirmatory trial, the investigators propose this multicenter preGallstep pilot trial.

The purpose of preGallstep is to assess the proportion of participants in the control group with complications in order to conduct more precise sample size estimation for a future pragmatic randomised clinical trial. Furthermore, the investigators want to assess the feasibility of implementing randomisation between different surgical techniques in a daily complex clinical setting.

Background In the Nordic countries, 80 to 200 surgical removals of the gallbladder (cholecystectomies) per 100000 inhabitants are performed annually making it one of the most common surgical procedures. In Denmark, over 7500 cholecystectomies are performed every year. Cholecystectomy is most often performed due to symptomatic gallstones in the gallbladder. However, common bile duct gallstones (CBDS) are found in 3.4% to 18% of patients undergoing cholecystectomy, with highest proportions during acute surgery. However, the most efficient and safest procedure to remove CBDS has yet to be identified.

A two-step approach including endoscopic retrograde cholangiography (ERC) with stone extraction and papillotomy with subsequent laparoscopic cholecystectomy has become the gold standard treatment for CBDS in Denmark. However, as the gallbladder is left in situ following successful clearance of CBDS there are high risks of symptom recurrence and gallstone complications.

ERC is an advanced endoscopic procedure and multiple ERCs are required in as much as 59% of patients. Temporary stents are placed in patients with failed stone clearance during ERC. This delays stone extraction and requires repeat-ERC. Acute pancreatitis is a feared complication following ERC and is reported to occur in 4% of patients (range 2.6% to 18%). Acute pancreatitis causes high mortality and morbidity and is associated with low long-term quality of life. Other long-term complications of ERC papillotomy include recurrent bile duct stones, cholangitis, stenosis, and an unknown risk of malignant transformation.

The most comprehensive study on gallstone disease included 34,200 unselected patients undergoing laparoscopic cholecystectomy and reported CBDS in 11.6% of which 16% were left untreated. In these 16%, one out of four patients experienced unfavourable outcomes such as complicated gallstone disease (pancreatitis, cholangitis, jaundice) or the need of ERC within 90 days. All other treatment strategies to remove CBDS caused lower risk of adverse events when compared to leaving CBDS untreated.

The treatment of CBDS is, therefore, recommended to include both clearance of CBDS and a cholecystectomy.

This one-step approach including laparoscopic common bile duct exploration with gallstoneclearance (LCBDE) plus laparoscopic cholecystectomy is an emerging minimal-invasive approach for CBDS. The one-step LCBDE plus laparoscopic cholecystectomy approach seems to cause less postoperative pancreatitis although no significant associations have been published yet.

A Cochrane review of five RCTs of the one-step versus the two-step approach with ERC first including 621 patients concluded that the two approaches were comparable regarding stone clearance, morbidity, and mortality. Newer RCTs have shown comparable stone clearance proportions and comparable occurrence of short-term postoperative complications and mortality between the two approaches.

The most recently published meta-analyses find that LCBDE versus ERC is superior in terms of safety (perioperative complications, conversion rate to other procedure), CBDS clearance rate, hospital stay, operative time, in hospital costs, and stones recurrence. Trial Sequential Analysis of the two approaches has been performed but due to the small sample sizes available, they were unable to make final conclusions on patient safety or CBDS removal efficiency. In order to explore what sample size was needed to make a final conclusion on patient safety, Trial Sequential Analysis including all known RCTs has been performed. The outcome of interest was adverse events defined by short-term postoperative complications as defined by the single studies. Intention-to-treat data were extracted where possible, however, some studies excluded randomised patients without CBDS at intraoperative cholangiography or patients that did not complete the protocolled treatments. Most trials randomised patients with only a clinical suspicion of CBDS and only few RCTs randomised patients with CBDS proven by MRCP or EUL. Through meta-analysis, the total proportion of adverse events was found to be 16% (102/649) in the two-step approach. Based on Trial Sequential Analyses, with a relative risk reduction 20%, α at 0.05, β at 0.10, a diversity of 0%, and when a two-sided test was used, the total sample size required was 5060 participants for adverse events. Previous trials already included 1302 participants and the trial sequential monitoring boundaries for superiority, inferiority, or futility have not been reached. The literature has, thereby, not yet identified the safest procedure or which treatment the patients prefer to remove CBDS. More research on patient safety, stone clearance, and patient-centred outcomes is needed.

Methods Trial design The preGallstep pilot is an investigator-initiated multicentre randomised parallel group, clinical, pilot trial with blinded outcome assessment at 90 days.

Randomisation Participants will be randomised at the allocation ratio 1:1. Web-based randomisation will be handled centrally at the Copenhagen Trial Unit (CTU) using a concealed computer-generated allocation sequence with a varying block size concealed from investigators. The allocation sequence will be stratified for trial site. A trial nurse will enroll and allocate participants.

Participant timeline Both acute and non-acute patients may enter. The physician in charge will offer enrolment to eligible patients. After enrolment, the participant will be randomised to one of the two treatment approaches.

Baseline data including quality of life survey will be established by the trial nurse.

The patient will receive the trial intervention or control intervention no later than one week after randomisation. Follow-up for immediate complications within first 24 postoperative hours will be performed by the trial nurse (follow-up day 1).

Blood samples including amylase will be drawn following the procedure. If no immediate complications occur, the patients will be discharged within 24 hours following the procedure. A 90-day clinical follow-up will be performed to assess outcomes. Registration of lost to follow-up and reasons will also be assessed here.

Blinding Blinding of participants and surgeons is not possible. Most of the outcomes are dependent on physician assessment. To have blinded outcome assessment, the trial nurse who has not been part of the surgical team and who is blinded to treatment allocation will perform the follow-up visits. Outcome will be assessed by a blinded outcome committee of three experts not associated with the trial or the participating departments.

Statistical plan and data analysis As this is a pilot trial, a formal sample size calculation is not necessary. A sample size of 150 participants is deemed feasible to include and randomised within 18 months, and it should be sufficient to base a formal size calculation on for the planning of a large pragmatic trial.

Statistical analysis will be performed according to the intention-to-treat principle. All patient included in the trial have CBDS according to the inclusion criteria and according to the best diagnostic modalities used in the clinic today (see above) and, therefore, the intention-to-treat principle can be used without any post-randomisation exclusions as done in some previous studies. Thereby, all patients with spontaneously passed stones at intra-operative cholangiography, lost-to follow up at 90 days, or patients not undergoing the full two-step procedures will be included in the statistical analyses. Analyses of the primary outcome will be performed for differences between intervention and control group after 90 days of follow-up. Dichotomous outcomes will be analysed using logistic regression. Continuous outcomes will be analysed using linear regression or van Eltern test. Analyses will be adjusted for the stratification variable. Odds ratios or mean differences will be reported with 95% confidence intervals and P-values. As this is a pilot trial, any significant result can be due to random errors and lack of power. It is therefore purely hypothesis generating.

Publications The investigators plan to publish a design article and an article describing the results of the preGallstep pilot trial. Furthermore, the results will be added to an updated meta-analysis. Authorship will be determined by the guidelines by the International Committee for Medical Journal Editors. Members of the trial steering committee as well as the principle investigator from each trial site will be invited as coauthors.

Collaborations The preGallstep trial is in collaboration between five major surgical departments in Denmark.

Investigators of each department have reached expert level of LC+LCBDE and have given consent of participation in the trial.

Protocol development, randomisation, data management, and surveillance of the trial are in collaboration with the Copenhagen Trial Unit (CTU). CTU is a non-specialty oriented clinical intervention research unit consisting of experienced trialists, clinicians, epidemiologists, statisticians, information-technology engineers, and information specialists.

Significance of the project There has not been a significant improvement to the treatment of bile stone disease since the introduction of laparoscopic surgery and ERC more than twenty years ago. Each year more than 750 new patients are diagnosed with CBDS in Denmark alone. ERC combined with LC is the treatment of choice but is affected by a high rate of severe complications and the risk of extended course of treatment.

The investigators propose a new method of treatment that might significantly reduce risk of complications, number of treatments needed, cost to society and improve patient satisfaction and make a difference to hundreds of people in Denmark alone each year.

Since this is a poorly researched area and large RCTs is needed it is important to make the necessary preparations by conducting a large pilot RCT

ELIGIBILITY:
Inclusion Criteria:

* Common bile duct stones identified by magnetic resonance cholangiopancreatography (MRCP).
* Age 18 years or older.
* Both interventions must be possible to perform within a clinically reasonable timeframe, as assessed by the investigator.
* Informed consent.

Exclusion Criteria:

Patients with acute cholangitis corresponding to a grade III (elevated serum bilirubin, fever, and/or elevated white blood cell count and signs of severe organ failure) according to Tokyo guidelines 2018 including severe organ failure.

* Common bile duct cysts shown by magnetic resonance cholangiopancreatography (MRCP), ultrasonography, computer tomography (CT), or cholangiography.
* Pancreatic/biliary/hepatic malignancies.
* Prior cholecystectomy or sphincterotomy.
* Chronic pancreatitis.
* If assessed by investigator that laparoscopic cholecystectomy is not possible, e.g. due to prior surgery or patient condition.
* Gastric bypass.
* Pregnancy confirmed by elevated choriogonadotropin (hCG) in women below 60 years.
* No informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications | 90 days
  Proportion of participants with postoperative complications corresponding to a Clavien-Dindo score of 2-5

SECONDARY OUTCOMES:
Stone clearance failure | perioperatively
  Rate of participants with incomplete stone clearance
Number of procedures | 90 days after initial procedure
  Total number of procedures for each participant during 90 days follow-up
Lenght of hospital stay | 90 days
  Total length of hospital stay for each participant
Stone size | Perioperatively
  Size of biggest common bile duct stone (mm)
Number of stones | perioperatively
  Number of common bile duct stones
Stone extraction pathway | perioperatively
  Is LCBDE transcystic or transcholedocal?
Stone extraction method | perioperatively
  Equipment used for stone extraction
Cholangiography | perioperatively
  Stones on perioperative cholangiography (yes/no)
Procedure time | From start of initial procedure until 90 days follow-up
  Total time spend on all procedures (minutes)
Conversion to open surgery | From start of initial procedure until 90 days follow-up
  Number of procedures converted to open surgery

OTHER OUTCOMES:
Quality of Life survey | 90 days
  QoL score (SF-36) at baseline and after 90 days follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive disease center, Bispebjerg Hospital, Copenhagen NV, Not in US/Canada, Denmark

IPD SHARING:
Plan to Share IPD: Yes
After the results have been published, we aim to make a depersonalised dataset publicly available on, e.g. clinicaltrials.gov, and/or the EU ZENODO database. The final choice will reflect which platform(s) that are compliant with current legislation at that time.
Supporting Information: Study Protocol, SAP
Time Frame: After publication

REFERENCES:
- [Background] Ryberg AA, Fitzgibbons RJ Jr, Tseng A, Maffi TR, Burr LJ, Doris PE. Abnormal cholangiograms during laparoscopic cholecystectomy. Is treatment always necessary? Surg Endosc. 1997 May;11(5):456-9. doi: 10.1007/s004649900389. PMID 9153174
- [Background] Sarli L, Pietra N, Franze A, Colla G, Costi R, Gobbi S, Trivelli M. Routine intravenous cholangiography, selective ERCP, and endoscopic treatment of bile duct stones before laparoscopic cholecystectomy. Gastrointest Endosc. 1999 Aug;50(2):200-8. doi: 10.1016/s0016-5107(99)70225-7. PMID 10425413
- [Background] Collins C, Maguire D, Ireland A, Fitzgerald E, O'Sullivan GC. A prospective study of common bile duct calculi in patients undergoing laparoscopic cholecystectomy: natural history of choledocholithiasis revisited. Ann Surg. 2004 Jan;239(1):28-33. doi: 10.1097/01.sla.0000103069.00170.9c. PMID 14685097
- [Background] Balandraud P, Biance N, Peycru T, Tardat E, Bonnet PM, Cazeres C, Hardwigsen J. Fortuitous discovery of common bile duct stones: results of a conservative strategy. Gastroenterol Clin Biol. 2008 Apr;32(4):408-12. doi: 10.1016/j.gcb.2008.02.023. Epub 2008 Apr 9. PMID 18403152
- [Background] Hammarstrom LE, Holmin T, Stridbeck H, Ihse I. Long-term follow-up of a prospective randomized study of endoscopic versus surgical treatment of bile duct calculi in patients with gallbladder in situ. Br J Surg. 1995 Nov;82(11):1516-21. doi: 10.1002/bjs.1800821121. PMID 8535807
- [Background] Targarona EM, Ayuso RM, Bordas JM, Ros E, Pros I, Martinez J, Teres J, Trias M. Randomised trial of endoscopic sphincterotomy with gallbladder left in situ versus open surgery for common bileduct calculi in high-risk patients. Lancet. 1996 Apr 6;347(9006):926-9. doi: 10.1016/s0140-6736(96)91413-0. PMID 8598755
- [Background] Boerma D, Rauws EA, Keulemans YC, Janssen IM, Bolwerk CJ, Timmer R, Boerma EJ, Obertop H, Huibregtse K, Gouma DJ. Wait-and-see policy or laparoscopic cholecystectomy after endoscopic sphincterotomy for bile-duct stones: a randomised trial. Lancet. 2002 Sep 7;360(9335):761-5. doi: 10.1016/S0140-6736(02)09896-3. PMID 12241833
- [Background] Frossard JL, Hadengue A, Amouyal G, Choury A, Marty O, Giostra E, Sivignon F, Sosa L, Amouyal P. Choledocholithiasis: a prospective study of spontaneous common bile duct stone migration. Gastrointest Endosc. 2000 Feb;51(2):175-9. doi: 10.1016/s0016-5107(00)70414-7. PMID 10650260
- [Background] Moller M, Gustafsson U, Rasmussen F, Persson G, Thorell A. Natural course vs interventions to clear common bile duct stones: data from the Swedish Registry for Gallstone Surgery and Endoscopic Retrograde Cholangiopancreatography (GallRiks). JAMA Surg. 2014 Oct;149(10):1008-13. doi: 10.1001/jamasurg.2014.249. PMID 25133326
- [Background] Coelho-Prabhu N, Shah ND, Van Houten H, Kamath PS, Baron TH. Endoscopic retrograde cholangiopancreatography: utilisation and outcomes in a 10-year population-based cohort. BMJ Open. 2013 May 31;3(5):e002689. doi: 10.1136/bmjopen-2013-002689. PMID 23793659
- [Background] Horiuchi A, Nakayama Y, Kajiyama M, Kato N, Kamijima T, Graham DY, Tanaka N. Biliary stenting in the management of large or multiple common bile duct stones. Gastrointest Endosc. 2010 Jun;71(7):1200-1203.e2. doi: 10.1016/j.gie.2009.12.055. Epub 2010 Apr 18. PMID 20400079
- [Background] Ding X, Zhang F, Wang Y. Risk factors for post-ERCP pancreatitis: A systematic review and meta-analysis. Surgeon. 2015 Aug;13(4):218-29. doi: 10.1016/j.surge.2014.11.005. Epub 2014 Dec 24. PMID 25547802
- [Background] Castoldi L, De Rai P, Zerbi A, Frulloni L, Uomo G, Gabbrielli A, Bassi C, Pezzilli R; ProInf-AISP (Progetto Informatizzato Pancreatite Acuta, Associazione Italiana per lo Studio del Pancreas) Study Group. Long term outcome of acute pancreatitis in Italy: results of a multicentre study. Dig Liver Dis. 2013 Oct;45(10):827-32. doi: 10.1016/j.dld.2013.03.012. Epub 2013 Jul 3. PMID 23831129
- [Background] Das SL, Singh PP, Phillips AR, Murphy R, Windsor JA, Petrov MS. Newly diagnosed diabetes mellitus after acute pancreatitis: a systematic review and meta-analysis. Gut. 2014 May;63(5):818-31. doi: 10.1136/gutjnl-2013-305062. Epub 2013 Aug 8. PMID 23929695
- [Background] Petrov MS, Shanbhag S, Chakraborty M, Phillips AR, Windsor JA. Organ failure and infection of pancreatic necrosis as determinants of mortality in patients with acute pancreatitis. Gastroenterology. 2010 Sep;139(3):813-20. doi: 10.1053/j.gastro.2010.06.010. Epub 2010 Jun 9. PMID 20540942
- [Background] Pendharkar SA, Salt K, Plank LD, Windsor JA, Petrov MS. Quality of life after acute pancreatitis: a systematic review and meta-analysis. Pancreas. 2014 Nov;43(8):1194-200. doi: 10.1097/MPA.0000000000000189. PMID 25333403
- [Background] Frimberger E. Long-term sequelae of endoscopic papillotomy. Endoscopy. 1998 Nov;30(9):A221-7. doi: 10.1055/s-2007-1001444. No abstract available. PMID 9932785
- [Background] Tanaka M, Takahata S, Konomi H, Matsunaga H, Yokohata K, Takeda T, Utsunomiya N, Ikeda S. Long-term consequence of endoscopic sphincterotomy for bile duct stones. Gastrointest Endosc. 1998 Nov;48(5):465-9. doi: 10.1016/s0016-5107(98)70086-0. PMID 9831833
- [Background] Hakamada K, Sasaki M, Endoh M, Itoh T, Morita T, Konn M. Late development of bile duct cancer after sphincteroplasty: a ten- to twenty-two-year follow-up study. Surgery. 1997 May;121(5):488-92. doi: 10.1016/s0039-6060(97)90101-x. PMID 9142145
- [Background] Thorlund K, Devereaux PJ, Wetterslev J, Guyatt G, Ioannidis JP, Thabane L, Gluud LL, Als-Nielsen B, Gluud C. Can trial sequential monitoring boundaries reduce spurious inferences from meta-analyses? Int J Epidemiol. 2009 Feb;38(1):276-86. doi: 10.1093/ije/dyn179. Epub 2008 Sep 29. PMID 18824467
- [Background] Wetterslev J, Jakobsen JC, Gluud C. Trial Sequential Analysis in systematic reviews with meta-analysis. BMC Med Res Methodol. 2017 Mar 6;17(1):39. doi: 10.1186/s12874-017-0315-7. PMID 28264661
- [Background] Wetterslev J, Thorlund K, Brok J, Gluud C. Estimating required information size by quantifying diversity in random-effects model meta-analyses. BMC Med Res Methodol. 2009 Dec 30;9:86. doi: 10.1186/1471-2288-9-86. PMID 20042080
- [Background] Jarvinen TL, Sihvonen R, Bhandari M, Sprague S, Malmivaara A, Paavola M, Schunemann HJ, Guyatt GH. Blinded interpretation of study results can feasibly and effectively diminish interpretation bias. J Clin Epidemiol. 2014 Jul;67(7):769-72. doi: 10.1016/j.jclinepi.2013.11.011. Epub 2014 Feb 20. PMID 24560088
- [Background] Miura F, Okamoto K, Takada T, Strasberg SM, Asbun HJ, Pitt HA, Gomi H, Solomkin JS, Schlossberg D, Han HS, Kim MH, Hwang TL, Chen MF, Huang WS, Kiriyama S, Itoi T, Garden OJ, Liau KH, Horiguchi A, Liu KH, Su CH, Gouma DJ, Belli G, Dervenis C, Jagannath P, Chan ACW, Lau WY, Endo I, Suzuki K, Yoon YS, de Santibanes E, Gimenez ME, Jonas E, Singh H, Honda G, Asai K, Mori Y, Wada K, Higuchi R, Watanabe M, Rikiyama T, Sata N, Kano N, Umezawa A, Mukai S, Tokumura H, Hata J, Kozaka K, Iwashita Y, Hibi T, Yokoe M, Kimura T, Kitano S, Inomata M, Hirata K, Sumiyama Y, Inui K, Yamamoto M. Tokyo Guidelines 2018: initial management of acute biliary infection and flowchart for acute cholangitis. J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):31-40. doi: 10.1002/jhbp.509. Epub 2018 Jan 8. PMID 28941329
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] ASGE Standards of Practice Committee; Buxbaum JL, Abbas Fehmi SM, Sultan S, Fishman DS, Qumseya BJ, Cortessis VK, Schilperoort H, Kysh L, Matsuoka L, Yachimski P, Agrawal D, Gurudu SR, Jamil LH, Jue TL, Khashab MA, Law JK, Lee JK, Naveed M, Sawhney MS, Thosani N, Yang J, Wani SB. ASGE guideline on the role of endoscopy in the evaluation and management of choledocholithiasis. Gastrointest Endosc. 2019 Jun;89(6):1075-1105.e15. doi: 10.1016/j.gie.2018.10.001. Epub 2019 Apr 9. PMID 30979521
- [Result] Dasari BV, Tan CJ, Gurusamy KS, Martin DJ, Kirk G, McKie L, Diamond T, Taylor MA. Surgical versus endoscopic treatment of bile duct stones. Cochrane Database Syst Rev. 2013 Dec 12;2013(12):CD003327. doi: 10.1002/14651858.CD003327.pub4. PMID 24338858
- [Result] Cuschieri A, Lezoche E, Morino M, Croce E, Lacy A, Toouli J, Faggioni A, Ribeiro VM, Jakimowicz J, Visa J, Hanna GB. E.A.E.S. multicenter prospective randomized trial comparing two-stage vs single-stage management of patients with gallstone disease and ductal calculi. Surg Endosc. 1999 Oct;13(10):952-7. doi: 10.1007/s004649901145. PMID 10526025
- [Result] Noble H, Tranter S, Chesworth T, Norton S, Thompson M. A randomized, clinical trial to compare endoscopic sphincterotomy and subsequent laparoscopic cholecystectomy with primary laparoscopic bile duct exploration during cholecystectomy in higher risk patients with choledocholithiasis. J Laparoendosc Adv Surg Tech A. 2009 Dec;19(6):713-20. doi: 10.1089/lap.2008.0428. PMID 19792866
- [Result] Bansal VK, Misra MC, Rajan K, Kilambi R, Kumar S, Krishna A, Kumar A, Pandav CS, Subramaniam R, Arora MK, Garg PK. Single-stage laparoscopic common bile duct exploration and cholecystectomy versus two-stage endoscopic stone extraction followed by laparoscopic cholecystectomy for patients with concomitant gallbladder stones and common bile duct stones: a randomized controlled trial. Surg Endosc. 2014 Mar;28(3):875-85. doi: 10.1007/s00464-013-3237-4. Epub 2013 Oct 26. PMID 24162138
- [Result] Ding G, Cai W, Qin M. Single-stage vs. two-stage management for concomitant gallstones and common bile duct stones: a prospective randomized trial with long-term follow-up. J Gastrointest Surg. 2014 May;18(5):947-51. doi: 10.1007/s11605-014-2467-7. Epub 2014 Feb 4. PMID 24493296
- [Result] Lv F, Zhang S, Ji M, Wang Y, Li P, Han W. Single-stage management with combined tri-endoscopic approach for concomitant cholecystolithiasis and choledocholithiasis. Surg Endosc. 2016 Dec;30(12):5615-5620. doi: 10.1007/s00464-016-4918-6. Epub 2016 Apr 28. PMID 27126621
- [Result] Koc B, Karahan S, Adas G, Tutal F, Guven H, Ozsoy A. Comparison of laparoscopic common bile duct exploration and endoscopic retrograde cholangiopancreatography plus laparoscopic cholecystectomy for choledocholithiasis: a prospective randomized study. Am J Surg. 2013 Oct;206(4):457-63. doi: 10.1016/j.amjsurg.2013.02.004. Epub 2013 Jul 17. PMID 23871320
- [Result] Sgourakis G, Karaliotas K. Laparoscopic common bile duct exploration and cholecystectomy versus endoscopic stone extraction and laparoscopic cholecystectomy for choledocholithiasis. A prospective randomized study. Minerva Chir. 2002 Aug;57(4):467-74. PMID 12145577
- [Result] Bansal VK, Misra MC, Garg P, Prabhu M. A prospective randomized trial comparing two-stage versus single-stage management of patients with gallstone disease and common bile duct stones. Surg Endosc. 2010 Aug;24(8):1986-9. doi: 10.1007/s00464-010-0891-7. Epub 2010 Feb 5. PMID 20135172
- [Result] Rogers SJ, Cello JP, Horn JK, Siperstein AE, Schecter WP, Campbell AR, Mackersie RC, Rodas A, Kreuwel HT, Harris HW. Prospective randomized trial of LC+LCBDE vs ERCP/S+LC for common bile duct stone disease. Arch Surg. 2010 Jan;145(1):28-33. doi: 10.1001/archsurg.2009.226. PMID 20083751
- [Result] Pan L, Chen M, Ji L, Zheng L, Yan P, Fang J, Zhang B, Cai X. The Safety and Efficacy of Laparoscopic Common Bile Duct Exploration Combined with Cholecystectomy for the Management of Cholecysto-choledocholithiasis: An Up-to-date Meta-analysis. Ann Surg. 2018 Aug;268(2):247-253. doi: 10.1097/SLA.0000000000002731. PMID 29533266
- [Result] Singh AN, Kilambi R. Single-stage laparoscopic common bile duct exploration and cholecystectomy versus two-stage endoscopic stone extraction followed by laparoscopic cholecystectomy for patients with gallbladder stones with common bile duct stones: systematic review and meta-analysis of randomized trials with trial sequential analysis. Surg Endosc. 2018 Sep;32(9):3763-3776. doi: 10.1007/s00464-018-6170-8. Epub 2018 Mar 30. PMID 29603004
- [Result] Ricci C, Pagano N, Taffurelli G, Pacilio CA, Migliori M, Bazzoli F, Casadei R, Minni F. Comparison of Efficacy and Safety of 4 Combinations of Laparoscopic and Intraoperative Techniques for Management of Gallstone Disease With Biliary Duct Calculi: A Systematic Review and Network Meta-analysis. JAMA Surg. 2018 Jul 18;153(7):e181167. doi: 10.1001/jamasurg.2018.1167. Epub 2018 Jul 18. PMID 29847616
- [Result] Barreras Gonzalez JE, Torres Pena R, Ruiz Torres J, Martinez Alfonso MA, Brizuela Quintanilla R, Morera Perez M. Endoscopic versus laparoscopic treatment for choledocholithiasis: a prospective randomized controlled trial. Endosc Int Open. 2016 Nov;4(11):E1188-E1193. doi: 10.1055/s-0042-116144. PMID 27857966
- [Derived] Kirkegaard-Klitbo A, Shabanzadeh DM, Olsen MH, Lindschou J, Gluud C, Sorensen LT. One-step laparoscopic cholecystectomy with common bile duct exploration and stone extraction versus two-step endoscopic retrograde cholangiography with stone extraction plus laparoscopic cholecystectomy for patients with common bile duct stones: a randomised feasibility and pilot clinical trial-the preGallStep trial. Pilot Feasibility Stud. 2023 Feb 6;9(1):21. doi: 10.1186/s40814-023-01251-z. PMID 36740708
- See also: Online only article — https://www.intechopen.com/books/advances-in-endoscopic-surgery/laparoscopic-one-stage-vs-endoscopic-plus-laparoscopic-management-of-common-bile-duct-stones-a-prosp